CLINICAL TRIAL: NCT01794819
Title: The Usefulness of Point-of-care-testing for C-reactive Protein in Lower Respiratory Tract Infection or Acute Cough
Brief Title: Usefulness of C-reactive Protein Testing in Acute Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRP-ARK-01/10
Record Dates: First submitted 2013-02-16; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Tract Infections
Keywords: antibiotics; primary care; radiology/radiography; respiratory tract infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-reactive protein test (Experimental): The C-reactive protein test was performed in the intervention group at both the first and second consultations.
  The Afinion test system (Axis Shield) was used, which provides results within 5 minutes and before treatment was determined. This test is based on solid-phase sandwich immunometric analysis. The measurement range in whole blood samples is 8-200 mg/L.
  Interventions: Device: C-reactive protein test

INTERVENTIONS:
Device: C-reactive protein test — Results provides within 5 minutes. This test is based on solid-phase sandwich immunometric analysis. The measurement range in whole blood samples is 8-200 mg/L.
  Other Names: The Afinion test system (Axis Shield)

SUMMARY:
The aim of this study is to evaluate the usefulness in Russian general practice of C-reactive protein testing in patients with acute cough or lower respiratory tract infections.

In addition to studying the effect of C-reactive protein testing on the prescription of antibiotics, the purpose is to find out whether the frequency of referral to radiography could be reduced.

DETAILED DESCRIPTION:
Eighteen general practitioners, from both urban and rural offices, were randomised into intervention and control groups. All registrations were made by general practitioners in their offices.

The case report form was similar to that used in the GRACE study (Genomics to combat Resistance against Antibiotics in Community-acquired lower respiratory tract infections in Europe (www.grace-lrti.org) describing symptoms, findings, and treatment in lower respiratory tract infections.

* The clinical examination included a chest examination and the axillary temperature.
* After the clinical examination, the general practitioners recorded their provisional diagnosis.
* Chest radiography was accessible for all patients.

The C-reactive protein test was performed in the intervention group at both the first and second consultations. The Afinion test system was used, which provides results within 5 minutes and before treatment was determined. This test is based on solid-phase sandwich immunometric analysis.

General practitioners could prescribe any treatment, including antibiotics and other drugs for the cough and additional medication if deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* patients with lower respiratory tract infections/acute cough (including acute bronchitis, pneumonia, and infectious exacerbations of chronic obstructive pulmonary disease or asthma),
* age 18 years or older,
* an illness of less than 28 days duration,
* first consultation for the illness episode,
* being seen in a physician's office,
* written consent to participate.

Exclusion Criteria:

* an inability to fill out study documentation,
* being previously included in the study,
* immunocompromised status (HIV patients, immunosuppressive treatment),
* ongoing treatment with oral corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
the antibiotic prescribing rate | within the first 2 weeks after first consultation

SECONDARY OUTCOMES:
referral to radiography | within the first 2 weeks after first consultation

OTHER OUTCOMES:
rate of recovery at the follow-up consultation | within the first 2 weeks after first consultation
  Rate of recovery at the follow-up consultation after 2 weeks with the following five alternatives: "fully recovered", "almost recovered", "slightly improved", "unchanged", and "worse". Consultations with the general practitioner within 2 weeks and complications (in need of hospitalisation) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hasse Melbye, PhD, Study Chair — University of Tromsø, Department of Community Medicine; Elena A Andreeva, MD, MPH, Principal Investigator — Northern State Medical University, Family Medicine Department
Locations (1):
- Northern State Medical University, Arkhangelsk, Russia

REFERENCES:
- [Derived] Smedemark SA, Aabenhus R, Llor C, Fournaise A, Olsen O, Jorgensen KJ. Biomarkers as point-of-care tests to guide prescription of antibiotics in people with acute respiratory infections in primary care. Cochrane Database Syst Rev. 2022 Oct 17;10(10):CD010130. doi: 10.1002/14651858.CD010130.pub3. PMID 36250577
- [Derived] Andreeva E, Melbye H. Usefulness of C-reactive protein testing in acute cough/respiratory tract infection: an open cluster-randomized clinical trial with C-reactive protein testing in the intervention group. BMC Fam Pract. 2014 May 2;15:80. doi: 10.1186/1471-2296-15-80. PMID 24886066